CLINICAL TRIAL: NCT00888095
Title: The Clinical Effect of Bilateral Deep Brain Stimulation of the Subthalamic Nucleus (STN-DBS) Versus Bilateral Deep Brain Stimulation of the Caudal Zona Incerta (cZI-DBS) in Patients With Idiopathic Parkinson's Disease
Brief Title: Deep Brain Stimulation (DBS) For Parkinson's Disease: Caudal Zona Incerta Versus Subthalamic Nucleus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Dr. A. Kupsch, Department of Neurology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DBS in the caudal Zona incerta
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Parkinson's Disease
Keywords: deep brain stimulation; caudal Zona incerta; Nucleus subthalamicus; Parkinson's disease; randomized; blinded; Movement disorder
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): caudal Zona incerta (cZI)
  Interventions: Procedure: deep brain stimulation
- 2 (Experimental): Nucleus subthalamicus (STN)
  Interventions: Procedure: deep brain stimulation

INTERVENTIONS:
Procedure: deep brain stimulation — electrode implantation in either STN or cZI

SUMMARY:
The aim of this study is to analyze the effects of two different targets of deep brain stimulation: caudal Zona incerta and Nucleus subthalamicus. The present study will investigate the effects of DBS using a blind, randomized and stratified design in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a severe neurological movement disorder comprising the triad of symptoms of bradykinesia, rigidity and tremor. It can be effectively treated with dopaminergic replacement therapy in the early course of the disease; however, after 5-10 years medical therapy is insufficient in the majority of patients. Since the early 90s the implantation of electrodes into the Nucleus subthalamicus (STN), (deep brain stimulation; DBS) has been established. DBS in PD- patients provides a definite and longlasting relief of motor symptoms and impaired quality of life compared to optimized medical treatment (Deuschl et al. 2006). Conventionally, electrodes are implanted into STN but other targets such as the pedunculopontine nucleus or the Zona incerta (ZI) have been reported to be useful. Importantly, the ZI has a key role in connection loops from the basal ganglia, thalamic regions and cortex. Retrospective studies of DBS-treated patients show relief of symptoms in DBS- treated PD patients, with the contacts of the electrodes being located to the ZI (Voges et al., 2002; Hamel et al., 2003a, 2003b). However, no prospective randomized studies analysing the effect of bilateral DBS comparing the targets of the caudal ZI (cZI) and STN are available. Therefore, the present study will investigate the effect and tolerance of DBS in both targets in a blind, randomized and stratified design in a total of 70 PD patients (see below for inclusion end exclusion criteria). The impairment of movement and quality of life will be assessed via established scales. Effects, tolerance and side effects of DBS will be monitored closely and re-assessed for a period of twelve months. Primary study criteria include UPDRS-III and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (criteria of the British Brain Bank: L-DOPA- or Apomorphin-sensitivity of more than 30% or typical Parkinsonian tremor while resting)
* duration of disease > 18 months
* age between 18 and 75 Jahren
* relevant disablement in daily activities/ impairment despite medical mental therapy
* informed and signed consent of the patient

Exclusion Criteria:

* major depression with suicidal thoughts (Becks Depressions Inventory-Score > 25); depressions in the past are no exclusion criterion
* Mattis Dementia Rating Scale-score < 130
* stereotactic brain operations in the past
* significant brain atrophy
* increased bleeding tendency
* reduced infection defense
* relevant cerebrovascular disease
* acute psychosis (benign and/or hallucinations in the past are no exclusion criterion)
* a physical and/or mental illness which is likely to affect the study procedures in a negative way (e.g., cancer with reduced life expectancy)
* abuse of drugs or alcohol
* female study participants of child- bearing age without adequate contraception
* women during pregnancy or lactation
* no sufficient knowledge of the German language to answer the questionnaires
* other surgical contraindications
* participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Improvement of scores (UPDRS III, PDQ-39) in Stim-ON and Med-OFF in a standard clinical check-up (CAPSIT) 12 and 24 months after operation compared to primary inclusion examination | 24 months

SECONDARY OUTCOMES:
Changes in dysarthria, other symptoms (subitems of UPDRS-III), dyskinesia (UPDRS-IV), impairment of gait, on-off fluctuations | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Kupsch, MD, Principal Investigator — Department of Neurology, Charité
Locations (1):
- Department of Neurology and Neurosurgery, Berlin, Germany

REFERENCES:
- [Background] Giladi N, Tal J, Azulay T, Rascol O, Brooks DJ, Melamed E, Oertel W, Poewe WH, Stocchi F, Tolosa E. Validation of the freezing of gait questionnaire in patients with Parkinson's disease. Mov Disord. 2009 Apr 15;24(5):655-61. doi: 10.1002/mds.21745. PMID 19127595